CLINICAL TRIAL: NCT02928939
Title: Therapeutic Conflicts in Hospitalized Patients: Retrospective Analyses of Patients With GI Bleeding or Exacerbated Diabetes and Impact of Multimorbidity.
Brief Title: Therapeutic Conflicts and Multimorbidity
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other); Center of Competence Multimorbidity, Zurich (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016-00525
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Gastrointestinal Hemorrhage; Diabetes Complications; Multimorbidity
Keywords: multimorbidity; multiple chronic conditions; drug-drug interactions; drug-disease interactions; polypharmacy; Oral anticoagulants; Steroids
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Diabetes Complications; Multiple Chronic Conditions | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Multimorbid patients
  Interventions: Other: drug-drug or drug-disease interaction

INTERVENTIONS:
Other: drug-drug or drug-disease interaction

SUMMARY:
Clinical practice guidelines do not take into account multimorbidity and various potential therapeutic conflicts. Identifying and quantifying therapeutic conflicts is crucial in multimorbid patients having more than two acute or chronic diseases. Guidance should be available for frequent encountered situations, e.g. gastrointestinal bleeding or exacerbation of diabetes mellitus.

DETAILED DESCRIPTION:
The study investigates multimorbidity in view of the occurrence of two different therapeutic conflicts or dilemma situations, respectively. The first concerns patients with diagnosis of gastrointestinal bleeding and prescription of anticoagulants or/and antiplatelet drugs (e.g., warfarin, clopidogrel and acetylsalicylic acid) as a risk factor for bleeding events. The second concerns patients with diagnosis of exacerbated diabetes mellitus and prescription of corticosteroids as a risk factor for worsening of blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at the University Hospital Zurich, USZ
* Male and female patients, aged 18 years or older
* Fulfilling the criteria for Use Case A or B (i.e. patients with gastrointestinal bleeding and anticoagulants or antiplatelet drugs, Use Case A or patients with diabetes mellitus and/or systemic corticosteroids, Use Case B)

Exclusion Criteria:

* If potential participants have a statement in the electronic medical record or elsewhere to refuse study participation, this represents exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We investigate in the field of multimorbidity in a tertiary hospital regarding therapeutic conflicts of GI bleeding and diabetes exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 1101 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Patients with gastrointestinal bleeding and anticoagulants or antiplatelet drugs | 5 years
  Do anticoagulants or antiplatelet drugs increase the risk of repeated bleeding in patients with gastrointestinal bleeding?
Patients with diabetes mellitus and systemic corticosteroids | 5 years
  Do systemic corticosteroids increase the risk of exacerbation in patients with diabetes mellitus?

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Battegay, Prof. MD, Study Director — University Hospital Zurich, Department of Internal Medicine; Klarissa Siebenhüner, MD, Principal Investigator — University Hospital Zurich, Department of Internal Medicine; Patrick Beeler, MD, Study Chair — University Hospital Zurich, Department of Internal Medicine
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided